CLINICAL TRIAL: NCT01008033
Title: Safety and Efficacy of Topical IDP-108 Versus Vehicle in Patients With Onychomycosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dow Pharmaceutical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DPSI-IDP-108-P3-01
Record Dates: First submitted 2009-11-03; First posted 2009-11-05 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- IDP-108 (Experimental)
  Interventions: Drug: IDP-108
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: IDP-108 — Topical application once a day for 48 weeks
  Arms: IDP-108
Drug: Vehicle — Topical application once a day for 48 weeks
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of topical application of IDP-108 versus vehicle in treating patients with onychomycosis.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed onychomycosis of the target nail
* Presence of mild to moderate onychomycosis, defined as 20 - 50% of the area of the target nail being clinically affected
* Has a positive KOH examination from the target nail
* Has a positive dermatophyte culture from the target nail

Exclusion Criteria:

* Presence of any disease or condition that might cause nail abnormalities or may interfere with the evaluation of the study drug
* Use of any systemic antifungal therapy within 4 weeks prior to the Screening visit or non-responsive to systemic antifungal therapy for onychomycosis
* Use of any prescription or over-the-counter topical antifungal therapy for the toenails within 4 weeks prior to the Screening visit
* Woman who is pregnant, nursing an infant, or planning a pregnancy during the study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Actual)
Dates: Start 2009-11; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who achieve clinical cure | 52 weeks

SECONDARY OUTCOMES:
Percentage of patients who achieve clinical efficacy | 52 weeks
Percentage of patients who achieve mycologic cure | 52 weeks

CONTACTS AND LOCATIONS:
Locations (72):
- United States (33):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - HOPE Research Institute, Phoenix, Arizona
  - Therapeutics Clinical Research, San Diego, California
  - University Clinical Trials, Inc, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Longmont Medical Research Network, Longmont, Colorado
  - The Savin Center, PC, New Haven, Connecticut
  - Foot and Ankle Associates of Florida, Inc, Altamonte Springs, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Ameriderm Research, Ormond Beach, Florida
  - Augusta Centre for Dermatology and Skin Renewal, LLC, Augusta, Georgia
  - Gwinnett Clinical Research Center, Inc., Snellville, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Hudson Dermatology, Evansville, Indiana
  - Dermatology Specialists, Louisville, Kentucky
  - Michigan Center for Research Corp., Clinton Township, Michigan
  - Academic Dermatology, Albuquerque, New Mexico
  - Impact Clinical Trials, New Hyde Park, New York
  - Radiant Research, Cinncinati, Ohio
  - Haber Dermatology & Cosmetic Surgery, South Euclid, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University School of Podiatric Medicine, Philadelphia, Pennsylvania
  - Palmetto Clinical Trial Services, LLC, Greenville, South Carolina
  - Rivergate Dermatology, Goodlettsville, Tennessee
  - Austin Dermatology Associates, Austin, Texas
  - J & S Studies, Inc., College Station, Texas
  - Baylor Research Institute, Dallas, Texas
  - Stephen Miller, MD, PA, San Antonio, Texas
  - Dermatology Resarch Center, Salt Lake City, Utah
  - The Education and Research Foundation, Inc., Lynchburg, Virginia
  - Virginia Clinical Research, Inc, Norfolk, Virginia
  - Aurora Advanced Healthcare, Inc. - Clinical Research Center, Milwaukee, Wisconsin
- Canada (7):
  - Kirk Barber Research, Calgary, Alberta
  - Stratica Medical, Edmonton, Alberta
  - Ultranova Skincare, Barrie, Ontario
  - Mediprobe Research, New London, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Centre de Recherche Dermatologique du Québec Métropolitain, Québec, Quebec
- Japan (32):
  - Kaken Investigational Site, Dazaifu, Fukuoka
  - Kaken Investigational Site - Chuo-ku #1, Fukuoka, Fukuoka
  - Kaken Investigational Site - Chuo-ku #2, Fukuoka, Fukuoka
  - Kaken Investigational Site - Higashi-ku, Fukuoka, Fukuoka
  - Kaken Investigational Site - Minami-ku #1, Fukuoka, Fukuoka
  - Kaken Investigational Site - Minami-ku #2, Fukuoka, Fukuoka
  - Kaken Investigational Site, Itoshima, Fukuoka
  - Kaken Investigational Site - Atsubetsu-ku #1, Sapporo, Hokkaido
  - Kaken Investigational Site - Atsubetsu-ku #2, Sapporo, Hokkaido
  - Kaken Investigational Site - Atsubetsu-ku #3, Sapporo, Hokkaido
  - Kaken Investigational Site - Chuo-ku, Sapporo, Hokkaido
  - Kaken Investigational Site - Kita-ku, Sapporo, Hokkaido
  - Kaken Investigational Site - Kiyota-ku, Sapporo, Hokkaido
  - Kaken Investigational Site - Nishi-ku, Sapporo, Hokkaido
  - Kaken Investigational Site - Shiroishi-ku, Sapporo, Hokkaido
  - Kaken Investigational Site - Teine-ku #1, Sapporo, Hokkaido
  - Kaken Investigational Site - Teine-ku #2, Sapporo, Hokkaido
  - Kaken Investigational Site, Kawasaki, Kanagawa
  - Kaken Investigational Site, Nagasaki, Nagasaki
  - Kaken Investigational Site, Ginowan, Okinawa
  - Kaken Investigational Site, Naha, Okinawa
  - Kaken Investigational Site, Nakagami, Okinawa
  - Kaken Investigational Site - Okinawa #1, Okinawa, Okinawa
  - Kaken Investigational Site - Okinawa #2, Okinawa, Okinawa
  - Kaken Investigational Site, Urasoe, Okinawa
  - Kaken Investigational Site, Kawaguchi, Saitama
  - Kaken Investigational Site - Nakano-ku #1, Nakano-ku, Tokyo
  - Kaken Investigational Site - Nakano-ku #2, Nakano-ku, Tokyo
  - Kaken Investigational Site - Setagaya-ku #1, Setagaya-ku, Tokyo
  - Kaken Investigational Site - Setagaya-ku #2, Setagaya-ku, Tokyo
  - Kaken Investigational Site - Shinagawa-ku #1, Shinagawa-ku, Tokyo
  - Kaken Investigational Site - Shinagawa-ku #2, Shinagawa-ku, Tokyo

REFERENCES:
- [Derived] Gupta AK, Elewski BE, Sugarman JL, Ieda C, Kawabata H, Kang R, Pillai R, Olin JT, Watanabe S. The efficacy and safety of efinaconazole 10% solution for treatment of mild to moderate onychomycosis: a pooled analysis of two phase 3 randomized trials. J Drugs Dermatol. 2014 Jul;13(7):815-20. PMID 25007364